CLINICAL TRIAL: NCT00383760
Title: A Phase II Study of the Halichondrin B Analog E7389 as Second Line Therapy for Patients With Locally Advanced Unresectable or Metastatic Pancreatic Cancer
Brief Title: Eribulin Mesylate as Second-Line Therapy for Locally Advanced, Unresectable, or Metastatic Pancreatic Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00173; PHL-049 (Other Grant/Funding Number: N01CM17107); CDR0000502291 (Other Grant/Funding Number: N01CM17107); N01CM62203 (NIH)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Adenocarcinoma of the Pancreas; Pancreatic Cancer; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (eribulin mesylate) (Experimental): Patients receive E7389 IV on days 1 and 8.
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog

SUMMARY:
This phase II trial is studying how well E7389 works as second-line therapy in treating patients with locally advanced, unresectable, or metastatic pancreatic cancer. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response (complete and partial) to E7389 in patients with locally advanced, unresectable, or metastatic pancreatic adenocarcinoma that progressed after prior gemcitabine hydrochloride-based therapy.

SECONDARY OBJECTIVE:

I. To determine the antitumor activity of E7389, in terms of median survival, 1-year survival rate, response or stable disease duration, toxicity, and time to disease progression, in these patients.

OUTLINE: This is an open-label, multicenter study. Patients receive eribulin mesylate IV on days 1 and 8. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, all patients are followed at 4 weeks. Patients with complete response, partial response, or stable disease are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed pancreatic carcinoma (locally advanced, unresectable or metastatic)
* measurable disease (at least 1 lesion accurately measured in at least 1 dimension (longest diameter as >20mm with conventional techniques or >10mm with spiral CT scan)
* >=4 weeks from any major surgery
* Up to 1 prior line of gemcitabine based systemic therapy (single agent/combination therapy) for locally advanced/metastatic disease with evidence of disease progression. Prior therapy with inhibitors of angiogenesis and/or the epidermal growth factor receptor permitted. Last chemotherapy dose >=4 weeks prior to randomization.
* May have received prior 5FU (+/- folinic acid)/gemcitabine given concurrently with radiation as a "radiation sensitizer". Last chemotherapy dose >=4 weeks prior to randomization.
* Prior radiation treatment >=4 weeks prior to randomization
* Age >18 years.
* Life expectancy >=3 months
* ECOG< 2(Karnofsky-60%)
* leukocytes>3,000/mcL
* absolute neutrophil count>1,500/mcL
* platelets>100,000/mcL
* total bilirubin < 1.5 UNL
* AST/ALT≤2.5x institutional ULN
* creatinine within institution limits OR creatinine clearance>60mL/min/1.73m2 for patients with creatinine levels above institution limits
* concurrent use of inhibitors/inducers of CYP3A4 are prohibited during the study treatment period
* effects of E7389 on developing human fetus are unknown. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand/willingness to sign written informed consent

Exclusion Criteria:

* chemotherapy/radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* May not be receiving other investigational agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to E7389
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study
* Pregnant women excluded because E7389 is an antitubulin agent with the potential for teratogenic/abortifacient effects
* HIV-positive patients on combination antiretroviral therapy are ineligible because of potential for p PK interactions with E7389
* Other active malignancies in past 5 years except for cervical carcinoma in situ and non-melanomatous skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Moore, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- E7389: Patients receive E7389 IV on days 1 and 8.
  eribulin mesylate: Given IV
Period: Overall Study
Arm/Group | E7389
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Eribulin Mesylate): Patients receive E7389 IV on days 1 and 8.
  eribulin mesylate: 1.4mg/m2 given IV weekly day 1,8 every 21 days (1 cycle).
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 62 [34 to 79]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Region of Enrollment [Number; unit: participants]
  Canada | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete and Partial) Evaluated Using RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
participants | 0

2. Secondary Outcome: Stable Disease Rate, Evaluated Using RECIST Criteria
Description: Stable disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
percentage of participants | 33 [15 to 59]

3. Secondary Outcome: Median Survival Time
Description: Estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
months | 6 [1 to 21]

4. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method.
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
percentage of participants | 58 [25 to 81]

5. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method.
Time Frame: At 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
participants | 0

6. Secondary Outcome: Median Time to Disease Progression
Description: Estimated using the Kaplan-Meier method.
Time Frame: Duration of time from start of treatment until the criteria for progression are met, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
months | 1.5 [1 to 9]

7. Secondary Outcome: Time to Progression
Description: Estimated using the Kaplan-Meier method.
  Median time to progression
Time Frame: At 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 15
months | 1.4 [1.2 to 8.5]

8. Secondary Outcome: Time to Progression
Description: Estimated using the Kaplan-Meier method.
Time Frame: At 1 year
Population: Time to progression at 1 year not analyzed
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 0

9. Secondary Outcome: Response Duration
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 3 years
Population: Data were not collected
Arm/Group | E7389
Number analyzed (Participants) | 0

10. Secondary Outcome: Toxicity
Description: Types of Gr 3 or greater adverse events that are atleast possibly related to study drug
Time Frame: All patients will be evaluable for toxicity from the time of their first treatment with E7389.
Measure: Number; unit: Types of adverse event
Arm/Group | E7389
Number analyzed (Participants) | 15
Types of adverse event | 8

11. Secondary Outcome: Objective Stable Disease Rate
Description: Objective stable disease rate Using RECIST
Time Frame: Upto 3 years
Population: Data was not collected
Arm/Group | E7389
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Eribulin Mesylate)
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Eribulin Mesylate) (N=15)
Dry skin (Skin and subcutaneous tissue disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Creatinine increased (Investigations) | 1
Death NOS (General disorders) | 2
Constipation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Eribulin Mesylate) (N=15)
Lymphocyte count decreased (Investigations) | 14
Abdominal pain (Gastrointestinal disorders) | 13
Anemia (Blood and lymphatic system disorders) | 13
Alkaline phosphatase increased (Investigations) | 12
Fatigue (General disorders) | 12
Nausea (Gastrointestinal disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Constipation (Gastrointestinal disorders) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 10
White blood cell decreased (Investigations) | 10
Alanine aminotransferase increased (Investigations) | 9
Neutrophil count decreased (Investigations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less